CLINICAL TRIAL: NCT01187043
Title: A Single-Blind, Placebo Run-in, Phase I/II Study Comparing Five Oral Doses of Proellex®
Brief Title: Determination of the Lowest, Safe and Effective Dose of Proellex
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZP-204
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-06

CONDITIONS: Amenorrhea
Keywords: Liver Function; Steady State Exposure
MeSH Terms: conditions — Amenorrhea | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ARM 1 (Experimental): 1 mg Proellex
  Interventions: Drug: Proellex
- ARM 2 (Experimental): 3 mg Proellex
  Interventions: Drug: Proellex
- ARM 3 (Experimental): 6 mg Proellex
  Interventions: Drug: Proellex
- ARM 4 (Experimental): 9 mg Proellex
  Interventions: Drug: Proellex
- ARM 5 (Experimental): 12 mg proellex
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — 1 capsule 1x/day of 1 mg(ARM1), 3 mg(ARM2), 6 mg(ARM3), 9 mg(ARM4) or 12 mg(ARM5)
  Other Names: CDB-4124; Telapristone acetate

SUMMARY:
The purpose of this study is to determine the effects of five different doses of Proellex on menses, ovulation, liver function, and steady state exposure in women of reproductive age.

DETAILED DESCRIPTION:
A phase I/II, 5 arm, single blind study, comparing five doses of Proellex to matching placebo in healthy adult female subjects of reproductive age. Exposure to study drug will be for up to 10 weeks. In-clinic pharmacokinetic (PK) assessments will be made on the first day of dosing and on the last day (week 10). Office visits will occur every week to assess liver function and trough blood concentrations for Proellex and primary metabolite. Daily vaginal bleeding diaries will be maintained during the course of the study. A single blind run-in period of up to 56 days will begin the study to assess baseline menstrual patterns will be utilized. Twelve subjects per treatment group (total 60 subjects) will be assigned to each dose. New groups will not begin dosing until the previous dose group has completed. Daily treatments will be either 1 mg, 3 mg, 6 mg, 9 mg, 12 mg Proellex. A single blind run-in period using placebo will be incorporated to establish baseline parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide a written informed consent.
* Healthy adult females between 18 and 50 years of age. Included in this group are women with the following conditions, not currently receiving drug treatment:

  * Excessive menstrual bleeding;
  * Menstrual pain;
  * Confirmed uterine fibroids; and
  * Confirmed endometriosis
* Normal menstrual cycle of 26-32 days
* Agree not to attempt to become pregnant
* Agree to limit alcohol consumption to no more than 2 drinks per week and to avoid alcohol consumption within 48 hours of each visit
* Ability to swallow gelatin capsules Ability to complete a daily subject diary
* Willing to discontinue hormonal contraceptives and consent to use of double barrier contraceptive techniques over the course of the study.
* Has a negative pregnancy test at the Screening and Baseline visits An exception for the pregnancy test requirement will be granted for subjects reporting surgical sterilization in medical history
* A Body Mass Index (BMI) between 18 and 39 inclusive
* Is available for all treatment and follow-up visits

Exclusion Criteria:

* Subject is a post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy
* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the 7 month study period
* Women with abnormal liver enzymes or liver disease.
* Subject previously participated in Proellex clinical trials: ZPE-201, ZPU-003, ZPU-301, ZPU-302, ZPU-303, ZPU-304, ZPU-305, and ZPU-307.
* Received an investigational drug in the 30 days prior to the screening for this study
* Women with a history of PCOS
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, DHEA or hormonal products for at least 2 weeks prior to screening and during the study.
* Use of oral contraceptives or hormone releasing IUDs in the preceding 30 days. Use of Depo-Provera® in the preceding 6 months.
* Women currently using narcotics
* Women currently taking cimetidine or spironolactone
* Clinically significant abnormal findings on screening examination or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Sterling, MD, Principal Investigator — ICON Development Solutions
Locations (1):
- ICON Devlopment Solutions, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4 | ARM 5
Started | 12 | 10 | 12 | 12 | 12
Completed | 11 | 10 | 8 | 12 | 10
Not Completed | 1 | 0 | 4 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Unable to make scheduled visits | 1 | 0 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4 | ARM 5 | Total
Number analyzed (Participants) | 12 | 10 | 12 | 12 | 12 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (7.8) | 38.5 (7.6) | 37.1 (8.6) | 34.4 (8.3) | 36.3 (7.0) | 36.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 12 | 12 | 12 | 58
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 12 | 12 | 12 | 58

OUTCOME MEASURES:

1. Primary Outcome: Induction Amenorrhea
Description: Induction of amenorrhea as determined by suppression of ovulation and/or menses, measured by using ovulation timing kits and daily diary for bleeding. Five doses will be compared in an escalating-dose, to independent groups, to a run-in placebo treatment period.
Time Frame: 10 weeks
Population: Per protocol: subjects who exhibited trough levels of proellex on at least 7 of the 10 weekly visits during the dosing period
Measure: Number; unit: participants
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4 | ARM 5
Number analyzed (Participants) | 2 | 9 | 7 | 10 | 7
participants | 2 | 9 | 6 | 8 | 6

ADVERSE EVENTS:
Time Frame: From first dose to one week post dosing (about 11 weeks).
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4 | ARM 5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 1/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 6/10 | 7/12 | 11/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (N=12) | ARM 2 (N=10) | ARM 3 (N=12) | ARM 4 (N=12) | ARM 5 (N=12)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Moderately differentiated invasive ductal carcinoma considered by Pi to be unlikely related to treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (N=12) | ARM 2 (N=10) | ARM 3 (N=12) | ARM 4 (N=12) | ARM 5 (N=12)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ear ache (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal cramps (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abcess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URI (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insect bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal PAP smear (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irregular menses (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Mittelschmertz (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Yeast infection (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Benign breast lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights